CLINICAL TRIAL: NCT00961402
Title: Efficacy of an Exercise Intervention for the Prevention of PostPartum Depression
Brief Title: The Effect of Exercise on Preventing PostPartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903S61462; R21MH085176 (NIH)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: PostPartum Depression
Keywords: Exercise; PostParum Depression
MeSH Terms: conditions — Depression, Postpartum; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wellness Control (Experimental): Participants will receive health and wellness information and no exercise information.
  Interventions: Behavioral: Wellness Control
- Exercise Intervention (Experimental): Intervention will include motivational telephone-based intervention to increase exercise to 5 days per week for 30 minutes or more each session.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Wellness Control — 6-month wellness control
  Arms: Wellness Control
Behavioral: Exercise Intervention — 6 month exercise intervention
  Arms: Exercise Intervention

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of an exercise intervention for the prevention of postpartum depression. If efficacious, our intervention could be disseminated in "real world settings" in an effort to prevent postpartum depression.

DETAILED DESCRIPTION:
Recent estimates indicate that approximately 10-15% of women giving birth experience depression during the postpartum period (Dietz et al., 2007; Gaven et al., 2005). Research indicates that psychological interventions are efficacious for treating postpartum depression (Dennis & Hodnett, 2007). However, it is important to also focus on the prevention of postpartum depression given many women do not seek treatment (Dennis & Chung-Lee, 2006) and those who do seek treatment may have already experienced negative consequences related to depression including cessation of breastfeeding and poor maternal-child bonding (Dennis & McQueen, 2007; Murray et al., 1999). Unfortunately, research indicates that psychological interventions are not efficacious in the prevention of postpartum depression among women at risk for postpartum depression (for a review see Dennis & Creedy, 2004). Consequently, there is a need to test new and innovative interventions for the prevention of postpartum depression. Exercise interventions have been shown to be effective for the treatment of depression among adults and therefore, this intervention may be efficacious in the prevention of postpartum depression. The purpose of the present pilot study is to examine the feasibility of recruiting and retaining participants at risk for postpartum depression for a randomized trial examining an exercise intervention for the prevention of postpartum depression. We will also examine the preliminary efficacy of the exercise intervention on the prevention of postpartum depression. Specifically, 120 sedentary, healthy pregnant women who have a history of at least one depressive episode and/or have a maternal family history of depression will be recruited from various ObGyn clinics, psychiatry clinics, and via advertisements. Once the potential participants receive healthcare provider consent to exercise (approximately two weeks following a vaginal delivery and four weeks following a c-section), participants will then be randomly assigned to either an exercise intervention or a health and wellness contact control condition. The exercise condition will consist of telephone-based counseling sessions designed to motivate postpartum women to become physically active. This theory-based intervention will be based on interventions shown to be effective in previous studies. The contact control condition will consist of scheduled telephone sessions with a health educator on issues related to health and wellness (e.g., stress reduction, sleep, nutrition). The specific aims of the study will be 1) to determine the feasibility of recruiting and retaining pregnant and postpartum women for an exercise intervention trial and 2) to determine the effect of a home-based behavioral exercise intervention on depression (as measured by the Structured Clinical Interview for DSM-IV Axis I Disorders; SCID-I and the PHQ-9) among postpartum women. Physical activity adherence will be assessed using the 7-Day Physical Activity Recall Interview (Blair et al., 1985) and accelerometers (i.e., an objective assessment of physical activity).

ELIGIBILITY:
Inclusion Criteria:

* We will recruit healthy, sedentary (defined as exercising 60 minutes or less per week) women who are at least 18 years of age and at least 28 weeks pregnant or less than one month postpartum (n=120). Participants will be required to obtain written consent from their healthcare provider to participate. This written consent will be obtained following delivery of the newborn. Participants will complete a telephone screening interview to assess eligibility. Current depressive episode will be assessed using the PHQ-9 (cut-off will be 10 or higher). As we have done in previous trials, we will have a protocol in place that deals with participants expressing suicidal ideation ranging from referring them to their healthcare provider and/or calling emergency assistance, depending on intent. To be included, participants must be willing to be randomly assigned to either of the two study arms. Additionally, participants will read and sign a consent form approved by the University of Minnesota and have all of their questions will be answered prior to participating.

Exclusion Criteria:

* No healthcare provider consent to participate
* Pre-existing hypertension or diabetes
* Current participation in exercise (defined as exercising 60 or more minutes per week)
* Currently enrolled in another exercise or weight management study
* Less than 18 years of age
* Another member of household participating in the study
* Unable to speak, comprehend, read, or write fluently in the English language
* Unable to walk for 30 minutes continuously
* Musculoskeletal problems such as arthritis, gout, osteoporosis, or back, hip or knee pain that may interfere with exercising
* Exercise-induced asthma
* Any condition that would make exercise unsafe or unwise
* Taking medication that interferes with heart rate response to exercise such as beta blockers
* Hospitalization for a psychiatric disorder in the past six months
* Current depressive episode and/or currently receiving antidepressant medication or psychotherapy for depression (those who are depressed and who are not in treatment will be referred to their physician or psychiatrist for follow-up care)

In addition to the initial exclusion criteria listed above, we will withdraw the exercise intervention and instruct the participant to contact their healthcare provider if the participant develops a medical issue in which exercise would be unsafe.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Lewis, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis BA, Gjerdingen D, Schuver K, Avery M, Marcus BH. The effect of sleep pattern changes on postpartum depressive symptoms. BMC Womens Health. 2018 Jan 9;18(1):12. doi: 10.1186/s12905-017-0496-6. PMID 29316912
- [Derived] Lewis BA, Billing L, Schuver K, Gjerdingen D, Avery M, Marcus BH. The relationship between employment status and depression symptomatology among women at risk for postpartum depression. Womens Health (Lond). 2017 Apr;13(1):3-9. doi: 10.1177/1745505717708475. Epub 2017 May 7. PMID 28480799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from January, 2010 through May, 2011 and follow-up assessments were completed by November, 2011. Participants were recruited via advertisements to the general public.
Pre-assignment Details: The major reason for why participants who consented but did not participate was that they failed to return our telephone calls after they had their baby or we were unable to obtain physician consent for them to participate.
Groups:
- Wellness Control: Participants will receive health and wellness information and no exercise information.
  Exercise: 6-month exercise intervention vs. wellness control
- Exercise: Intervention will include motivational telephone-based intervention to increase exercise to 5 days per week for 30 minutes or more each session.
  Exercise: 6-month exercise intervention vs. wellness control
Period: Overall Study
Arm/Group | Wellness Control | Exercise
Started | 64 | 66
Randomized | 64 | 66
Completed | 63 | 61
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellness Control | Exercise | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.39 (4.63) | 31.69 (5.27) | 31.54 (4.95)
Sex/Gender, Customized [Number; unit: participants]
  Females | 64 | 66 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 61 | 64 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 55 | 55 | 110
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 64 | 66 | 130
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — This scale measures the participant's perception of stress. This is a 14 item scale ranging from 0-56, with higher scores indicating higher stress.
  units on a scale | 24.73 (6.98) | 23.21 (7.94) | 23.96 (7.50)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — This measure assess depressive symptoms. There are 9 items and scores range from 0-27 with higher scores indicating higher levels of depression.
  units on a scale | 6.56 (4.27) | 5.42 (3.28) | 5.99 (3.83)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — This measure assesses sleep problems. This 9-item measure ranges from 0-21 with higher scores indicating more sleep problems.
  units on a scale | 7.11 (3.08) | 7.11 (2.61) | 7.11 (2.84)

OUTCOME MEASURES:

1. Primary Outcome: Structured Clinical Interview for DSM-IV Axis I Disorders
Description: This measure was used to determine if participants met the diagnostic criteria for postpartum depression. This is a yes/no diagnostic tool and our data indicate percentage who meet criteria for depression.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Wellness Control | Exercise
Number analyzed (Participants) | 63 | 61
percentage of participants | 7.94 | 8.20

2. Secondary Outcome: 7-Day Physical Activity Recall Interview
Description: Physical activity during previous 7 days. This measure does not have a range given it is directly dependent upon number of minutes of physical activity per week. The intensity ranges from moderate (similar to a brisk walk), hard (similar to a jog), and very hard (similar to a run).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of physical activity minutes
Arm/Group | Wellness Control | Exercise
Number analyzed (Participants) | 63 | 61
Number of physical activity minutes | 123.3 (111.4) | 129.8 (87.5)

3. Secondary Outcome: Edinburgh Postnatal Depression Scale
Description: This scale is a continuous measure of postpartum depression. Range is 0-30 and a score of 10 or above may be considered depressed. Higher scores indicate higher depression.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Wellness Control | Exercise
Number analyzed (Participants) | 63 | 61
Score on a scale | 7.02 (4.64) | 4.69 (3.89)

4. Secondary Outcome: PHQ-9
Description: Continuous measure of depression. Scoring is on a scale of 0-27 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Wellness Control | Exercise
Number analyzed (Participants) | 63 | 61
Score on a scale | 5.22 (4.59) | 3.08 (3.04)

ADVERSE EVENTS:
Arm/Group | Wellness Control | Exercise
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66
Other Adverse Events (participants affected / at risk) | 0/130 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No